CLINICAL TRIAL: NCT01016015
Title: A Phase 2 Study of Temsirolimus (CCI-779, NSC 683864) and IGF-1 Receptor Antibody Cixutumumab (IMC-A12, NSC 742460) in Patients With Metastatic Sarcomas
Brief Title: Temsirolimus and Cixutumumab in Treating Patients With Locally Advanced, Metastatic, or Recurrent Soft Tissue Sarcoma or Bone Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01408; NCI-2011-01408 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000659358; 09-097 (Other: Memorial Sloan-Kettering Cancer Center); 8121 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00071 (NIH); N01CM00100 (NIH); P30CA008748 (NIH)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2014-05

CONDITIONS: Metastatic Osteosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Osteosarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Osteosarcoma; Sarcoma | interventions — cixutumumab; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cixutumumab and temsirolimus) (Experimental): Patients receive cixutumumab IV over 60 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cixutumumab; Other: Laboratory Biomarker Analysis; Drug: Temsirolimus

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase II trial studies how well temsirolimus and cixutumumab works in treating patients with locally advanced, metastatic, or recurrent soft tissue sarcoma or bone sarcoma. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cixutumumab, can block tumor growth by blocking the ability of tumor cells to grow and spread. Giving temsirolimus with cixutumumab may be an effective treatment for soft tissue or bone sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients progression-free at 12 weeks (progression free survival [PFS], defined as Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 complete response [CR] + partial response [PR] + stable disease [SD]) with (A) Insulin-like growth factor (IGF)-1receptor (R)+ soft tissue sarcomas; (B) IGF-1R+ bone tumors; or (C) IGF-1R(-) sarcomas, who are treated weekly with intravenous A12 (cixutumumab) and temsirolimus.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (defined as CR + PR). II. To determine the overall survival. III. To determine the correlation of clinical outcome with pre- and post-treatment IGF-1R pathway related markers in plasma (pre and post therapy), archived tissue, and pre- and post-treatment tumor biopsies.

OUTLINE:

Patients receive cixutumumab intravenously (IV) over 60 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed sarcoma of soft tissue or bone; all patients will have IGF-1R testing at Memorial Sloan-Kettering Cancer Center (MSKCC) by immunohistochemistry (IHC); patients with confirmation of IGF-1R status in pre-existing tumor specimens will be enrolled on one of three arms of the study:

  * Arm A: IHC IGF-1R (+) sarcomas of soft tissue
  * Arm B: IHC IGF-1R (+) sarcomas of bone
  * Arm C: Any IGF-1R (-) sarcomas
* Subjects must have metastatic and/or locally advanced or locally recurrent disease
* Patients treated at Memorial Sloan Kettering Cancer Center must consent to tumor biopsies before therapy and after the 2nd week of therapy; subjects who do not have accessible tumor for biopsy may be enrolled at the discretion of the Principal Investigator
* Patients must have measurable disease by RECIST 1.1; measurable disease (a 'target' lesion) is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT) (CT scan slice thickness no greater than 5 mm); >= 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable); and >= 20 mm by chest x-ray
* A minimum of 1 and a maximum of 4 prior systemic therapy regimens for recurrent/metastatic disease; the last dose of systemic therapy (include tyrosine kinase inhibitors) must have been given at least 4 weeks prior to initiation of therapy; patients receiving carmustine (BCNU) or mitomycin C must have received their last dose of such therapy at least 6 weeks prior to initiation of therapy
* Patients with brain metastasis that have been treated with definitive surgery or radiation and have been clinically stable for 3 months following the procedure with no neurological signs or symptoms and no requirement for systemic glucocorticoids are eligible for study
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count >= 1.5 x 10^9/l; patients with neutropenia on a familial basis may still be enrolled on study; please contact the Principal Investigator (PI) who will discuss the patient with Cancer Therapy Evaluation Program (CTEP)
* Platelets >= 100 x 10^9/l
* Total bilirubin =< 1.5 x upper limit of normal (ULN); in patients with bilirubin > 1-1.5 X ULN, the starting dose of temsirolimus is 15 mg/week
* Albumin >= 3 g/dL
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3.0 x institution ULN; in patients with ALT or AST elevated > 1.0- 3.0 X ULN, the starting dose of temsirolimus is 15 mg/week
* Serum creatinine =< 1.5 x ULN
* Serum glucose =< 120 mg/dL; nonfasting or fasting; if a patient has a non-fasting glucose of over 120 mg/dL, the patient may be retested in the fasting state to determine if they are eligible for study; a non-fasting glucose of 120 or less renders the patient eligible for study
* Fasting total cholesterol =< 300 mg/dL
* Fasting triglycerides =< 300 mg/dL; patients with neutropenia on a familial basis may still be enrolled on study; please contact the PI who will discuss the patient with CTEP
* Patients must not have current evidence of another malignancy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) and have pregnancy testing prior to study entry and for the duration of study participation (every 2 cycles of therapy); should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Adverse events related to prior tumor-specific therapy must have resolved to less than or equal to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version 4.0) grade 1 prior to study entry (except alopecia)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had major surgery or a course of glucocorticoid therapy lasting longer than 5 days within 4 weeks prior to entering the study, or those who have not recovered from adverse events to =< NCI CTCAE (version 4.0) grade 1, associated with surgery; excluded from such considerations are surgical changes not expected to improve, e.g. removal of muscle tissue; patients may be on replacement glucocorticoids for pre-existing glucocorticoid deficiency (e.g. Addison's disease) or topical glucocorticoids for dermatological conditions (e.g. psoriasis)
* Patients must be >= 4 weeks beyond treatment of any systemic therapy, other investigational therapy, biological, targeted agents or radiotherapy, and must have recovered to =< Grade 1 toxicity or previous baseline for each toxicity; specifically excluded are the laboratory examinations serum lipase or amylase (without overt pancreatitis), hypophosphatemia, hypomagnesemia, and lymphopenia; patients may have received palliative low dose radiotherapy to the limbs 1-4 weeks before this therapy provided pelvis, sternum, scapulae, vertebrae, or skull were not included in the radiotherapy field
* Patients may not have received prior IGFR1 inhibitors
* Patients may not have received prior mammalian target of rapamycin (mTOR) inhibitors (such as sirolimus, everolimus, ridaforolimus, or temsirolimus)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temsirolimus, A12, or other agents used in the study
* Patients with hyperglycemia, defined as fasting serum glucose above 120 mg/dl, or those patients already on oral anti-diabetic or insulin therapy
* Uncontrolled intercurrent illness including, but not limited to, known ongoing or active infection, including human immunodeficiency virus (HIV), active hepatitis B or C, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (specifically, atrial fibrillation or ventricular dysrhythmias except ventricular premature contractions), or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women and women who are breast-feeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2009-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tap, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (24):
- United States (22):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SUNY College at Old Westbury, Old Westbury, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Schwartz GK, Tap WD, Qin LX, Livingston MB, Undevia SD, Chmielowski B, Agulnik M, Schuetze SM, Reed DR, Okuno SH, Ludwig JA, Keedy V, Rietschel P, Kraft AS, Adkins D, Van Tine BA, Brockstein B, Yim V, Bitas C, Abdullah A, Antonescu CR, Condy M, Dickson MA, Vasudeva SD, Ho AL, Doyle LA, Chen HX, Maki RG. Cixutumumab and temsirolimus for patients with bone and soft-tissue sarcoma: a multicentre, open-label, phase 2 trial. Lancet Oncol. 2013 Apr;14(4):371-82. doi: 10.1016/S1470-2045(13)70049-4. Epub 2013 Mar 8. PMID 23477833

RESULTS

PARTICIPANT FLOW:
Groups:
- Cixutumumab and Temsirolimus: Patients receive cixutumumab IV over 60 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cixutumumab and Temsirolimus
Started | 178
Completed | 159
Not Completed | 19
Not completed — Not Treated | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 15

BASELINE CHARACTERISTICS:
Arm/Group | Cixutumumab and Temsirolimus
Number analyzed (Participants) | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 144
  >=65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 98
Region of Enrollment [Number; unit: participants]
  United States | 178

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate, Defined as CR + PR + SD, as Assessed by RECIST Criteria
Description: From study entry until recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurement recorded on study), death or date of last contact, assessed at 12 weeks
Time Frame: From study entry until recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurement recorded on study), death or date of last contact, assessed at 12 weeks
Measure: Number; unit: participants
Arm/Group | Cixutumumab and Temsirolimus
Number analyzed (Participants) | 159
participants
  Partial Response | 4
  Progression of Disease | 57
  Stable Disease | 98

ADVERSE EVENTS:
Arm/Group | Cixutumumab and Temsirolimus
Serious Adverse Events (participants affected / at risk) | 83/175
Other Adverse Events (participants affected / at risk) | 62/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cixutumumab and Temsirolimus (N=175)
Abdominal pain (Gastrointestinal disorders) | 3 (6)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood and lymph system disorder (Blood and lymphatic system disorders) | 1 (1)
Blood Bilirubin increase (Investigations) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3)
Colonic fistula (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Death NOS (General disorders) | 11 (11)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 9 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Edema-Limb (General disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hepatobiliary disorder (Hepatobiliary disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 7 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection and Infestations (Infections and infestations) | 3 (3)
Intracranial hemorrhage (Nervous system disorders) | 1 (2)
Localized edema (General disorders) | 1 (1)
Lung Infection (Infections and infestations) | 7 (8)
Lymphocyte count decrease (Investigations) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (2)
Mucositis-Oral (Gastrointestinal disorders) | 12 (14)
Muscle weakness lower limbs (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Paronychia (Infections and infestations) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2)
Platelet count decreased (Investigations) | 10 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorder (Renal and urinary disorders) | 3 (3)
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (7)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 7 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cixutumumab and Temsirolimus (N=175)
Activated partial thromboplastin time prolonged (Investigations) | 14 (25)
Alanine aminotransferase (Investigations) | 32 (60)
Alkaline phosphatase increased (Investigations) | 32 (175)
Aspartate aminotransferase increased (Investigations) | 31 (132)
Blood Bilirubin increased (Investigations) | 12 (29)
Cholesterol, High (Investigations) | 41 (139)
Creatinine increased (Investigations) | 19 (192)
Hyperglycemia (Metabolism and nutrition disorders) | 61 (915)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (21)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 40 (159)
Hypoalbuminemia (Metabolism and nutrition disorders) | 51 (509)
Hypocalcemia (Metabolism and nutrition disorders) | 26 (157)
Hypokalemia (Metabolism and nutrition disorders) | 15 (57)
Hyponatremia (Investigations) | 30 (133)
Hypophosphatemia (Metabolism and nutrition disorders) | 19 (52)
INR increased (Metabolism and nutrition disorders) | 31 (107)
Lymphocyte count decrease (Investigations) | 18 (98)
Neutrophil count decrease (Investigations) | 21 (59)
Platelet Count decrease (Investigations) | 50 (404)
White blood cell decrease (Investigations) | 44 (285)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less